CLINICAL TRIAL: NCT06744868
Title: A Single- and Multiple-Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of THDBH120 Injection in Healthy Subjects: A Randomized, Bouble-Blind, Placebo-Controlled Phase I Trial
Brief Title: A Single- and Multiple-Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of THDBH120 Injection in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tonghua Dongbao Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: THDBH120L101
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Healthy
MeSH Terms: interventions — Sagittal Abdominal Diameter; mycophenolic adenine dinucleotide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- THDBH120 injection (SAD) (Experimental)
  Interventions: Drug: THDBH120 injection (SAD)
- Placebo of THDBH120 injection (SAD) (Placebo Comparator)
  Interventions: Drug: Placebo of THDBH120 injection (SAD)
- THDBH120 injection (MAD) (Experimental)
  Interventions: Drug: THDBH120 injection (MAD)
- Placebo of THDBH120 injection (MAD) (Placebo Comparator)
  Interventions: Drug: Placebo of THDBH120 injection (MAD)

INTERVENTIONS:
Drug: THDBH120 injection (SAD) — Participants received escalating single doses of THDBH120 by subcutaneous injection.
  Arms: THDBH120 injection (SAD)
Drug: Placebo of THDBH120 injection (SAD) — Participants received single dose of placebo by subcutaneous injection.
  Arms: Placebo of THDBH120 injection (SAD)
Drug: THDBH120 injection (MAD) — Participants received multiple doses of THDBH120 once weekly for four weeks by subcutaneous injection.
  Arms: THDBH120 injection (MAD)
Drug: Placebo of THDBH120 injection (MAD) — Participants received placebo once weekly for four weeks by subcutaneous injection.
  Arms: Placebo of THDBH120 injection (MAD)

SUMMARY:
This study includes single-ascending dose cohorts (SAD cohorts) and multiple-ascending dose cohorts (MAD cohorts). The aim of this trial is to investigate the safety, tolerability, pharmacokinetics, and pharmacodynamics of THDBH120 injection in healthy patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Chinese subjects aged 18 to 45 years (inclusive), male or female;
* Body Mass Index (BMI) ≥ 19 kg/m2 and ≤ 28kg/m2, male weight ≥ 50 kg, females weight≥ 45 kg;
* Normal or abnormal but not clinically significant physical examination and vital signs at screening.

Exclusion Criteria:

* Have a diagnosis of type 2 diabetes or have had episode of severe hypoglycemia;
* Pulse rate is less than 50 bpm or more than 100 bpm at screening;
* 12-lead electrocardiogram with prolonged QTcF (male >450 ms, female >470 ms) or PR>200ms. Or any other situation in which a 12-lead ECG suggests a risk of ineligibility at screening;
* A history of pancreatitis (including chronic pancreatitis or idiopathic acute pancreatitis), abnormal amylase and lipase with clinical significance or gastrointestinal injury (e.g., chronic gastritis, peptic ulcer, recurrent gastroesophageal reflux disease, cholecystitis, and gallstones) or any gastrointestinal disease that interferes with gastric emptying (e.g., gastric bypass surgery, pyloric stenosis);
* Have a personal or family history of medullary thyroid carcinoma or have multiple endocrine neoplasia syndrome type 2;
* Use of SGLT inhibitors, DPP4 inhibitors, GLP-1 analogs, GLP-1 receptor agonists, and other drugs that investigators recognize may affect the study during the 3 months prior to randomization;
* Have had a significant change in weight during the 6 months prior to screening, such as weight loss > 10%, or recent significant changes in diet or exercise habits.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2023-12-19 (Actual); Primary Completion 2024-09-22 (Actual); Study Completion 2024-09-22 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Adverse Event(s) and Serious Adverse Event(s) | From the first drug administration to the follow-up visit (57 days after the last drug administration)

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of THDBH120. | Day 1 Pre-dose through Day 42 (SAD), Day 1 Pre-dose through Day 29 (MAD)
Pharmacokinetics (PK): Maximum Drug Concentration (Cmax) of THDBH120 | Day 1 Pre-dose through Day 42 (SAD), Day 1 Pre-dose through Day 29 (MAD)
Evaluate the Fasting Blood Glucose (FBG ) of THDBH120 | Day 1 Pre-dose through Day 8 (SAD), Day 1 Pre-dose through Day 29 (MAD)
Number of Participants With Anti-THBHD120 Antibodies | From the first drug administration to the follow-up visit (57 days after the last drug administration)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No